CLINICAL TRIAL: NCT04049760
Title: A Long-term, Open-label Study to Evaluate the Safety, Pharmacodynamics, and Efficacy of Migalastat in Subjects > 12 Years of Age With Fabry Disease and Amenable GLA Variants
Brief Title: Safety, Pharmacodynamics, and Efficacy of Migalastat in Pediatric Subjects (Aged >12 Years) With Fabry Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT1001-036; 2019-000222-21 (EudraCT Number)
Record Dates: First submitted 2019-07-30; First posted 2019-08-08 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Fabry Disease
Keywords: Lysosomal disease; migalastat
MeSH Terms: conditions — Fabry Disease | interventions — migalastat; larazotide acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- migalastat HCl 150 mg (Experimental): One migalastat 123 mg capsule equivalent to 150 mg migalastat HCl will be administered every other day (QOD) during the treatment period.
  Interventions: Drug: migalastat HCl 150 mg

INTERVENTIONS:
Drug: migalastat HCl 150 mg — migalastat HCl 150 mg capsule
  Other Names: migalastat; AT1001

SUMMARY:
This is a long-term, Open-label Study to Evaluate the Safety, Pharmacodynamics, and Efficacy of Migalastat in Subjects > 12 Years of Age With Fabry Disease and Amenable GLA Variants

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects diagnosed with Fabry disease > 12 years of age who completed Study AT1001-020
* Subject's parent or legally-authorized representative is willing and able to provide written informed consent and authorization for use and disclosure of personal health information or research-related health information, and subject provides assent, if applicable
* If of reproductive potential, both male and female subjects agreed to use a medically accepted method of contraception throughout the duration of the study and for up to 30 days after their last dose of migalastat

Exclusion Criteria:

* Subject's last available estimated glomerular filtration rate (eGFR) in the previous study was < 60 mL/min/1.73 m2
* Subject had advanced kidney disease requiring dialysis or kidney transplantation
* Subject received any investigational/experimental drug, biologic, or device within 30 days before baseline, with the exception of migalastat
* Subject anticipated starting gene therapy during the study period
* Subject had any intercurrent illness or condition at Visit 1 that may have precluded the subject from fulfilling the protocol requirements or suggested to the investigator that the potential subject may have an unacceptable risk by participating in this study
* Subject had a history of allergy or sensitivity to migalastat (including excipients) or other iminosugars (eg, miglustat, miglitol)
* Subject required treatment with Replagal® (agalsidase alfa) or Fabrazyme® (agalsidase beta)
* Subject required treatment with Glyset® (miglitol) or Zavesca® (miglustat)
* Female subject was pregnant or breast-feeding, or was planning to become pregnant during the study period
* In the opinion of the investigator, the subject and/or parent or legally-authorized representative was unlikely or unable to comply with the study requirements

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - University of South Florida, Tampa, Florida
  - The Emory Clinic, Atlanta, Georgia
  - University of Minnesota Masonic Children's Hospital and Clinics, Minneapolis, Minnesota
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Lysosomal & Rare Disorders Research & Treatment Center, Fairfax, Virginia
- Royal Free London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Migalastat HCl 150 mg: One migalastat 123 mg capsule (equivalent to 150 mg migalastat HCl) administered every other day (QOD) during the treatment period.
Period: Overall Study
Arm/Group | Migalastat HCl 150 mg
Started | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 16
Age, Customized [Count of Participants; unit: Participants]
  12 to < 16 years | 7
  16 to < 18 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 1
  Unknown or Not Reported | 0
Prior Enzyme Replacement Therapy (ERT) status [Count of Participants; unit: Participants]
  ERT-experienced | 8
  ERT-naive | 8

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and AEs (Adverse Events) Leading to Discontinuation of Study Drug
Description: Number of subjects with TEAE, SAE, and AE leading to discontinuation during the study period
Time Frame: Entire study
Measure: Count of Participants; unit: Participants
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 16
Participants
  Number of subjects with TEAEs | 13
  Number of subjects with SAE | 1
  Number of subjects with AE leading to discontinuation | 0

2. Secondary Outcome: Change From Baseline to Month 24 in Estimated Glomerular Filtration Rate (eGFR)
Description: Estimated GFR was calculated using the modified Schwartz formula according to the standards of the central laboratory.
Time Frame: Baseline, Month 24
Population: 8 subjects had eGFR calculated at Month 24 visit
Measure: Mean (Standard Deviation); unit: mL/min x 1.73 m2
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 8
mL/min x 1.73 m2 | -27.6 (8.88)

3. Secondary Outcome: Change From Baseline to Month 24 in Urine Protein Levels
Description: Renal function was assessed by urine protein levels (mg/L). Urine samples were collected as part of urinalysis.
Time Frame: Baseline, Month 24
Population: 7 subjects had urine protein value at Month 24
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 7
mg/L | 38.6 (79.03)

4. Secondary Outcome: Change From Baseline to Month 24 in Urine Albumin
Description: Renal function was assessed by urine albumin levels (mg/L). Urine samples were collected as part of urinalysis
Time Frame: Baseline, Month 24
Population: 6 subjects had urine albumin result at Month 24
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 6
mg/L | -12.7 (21.73)

5. Secondary Outcome: Change From Baseline to Month 24 in Left Ventricular Mass Index (LVMi)
Description: LVMi was assessed as a measure of cardiac impairment in the study participants. LVMi values for both M-mode and 2D views are presented.
Time Frame: Baseline, Month 24
Population: 8 subjects had LVMi results at Month 24
Measure: Mean (Standard Deviation); unit: g/m2
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 8
g/m2
  2D-mode View | 4.75 (16.679)
  M-mode View | 6.01 (9.014)

6. Secondary Outcome: Change From Baseline to Month 24 in Pediatric and Quality of Life Inventory™ (PedsQL™) Scores
Description: The Pediatric Quality of Life Inventory (PedsQL™) was a modular approach to measuring health-related quality of life (QoL) in healthy children and adolescents and those with acute and chronic health conditions. All components of the PedsQL were scored based on a scale of 0 (never) to 4 (almost always) and linearly transformed to a 0 to 100 scale as follows: 0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0. Psychosocial, physical, and total scores were calculated based on the response to the questions within the patient reported outcome. The psychosocial score for the PedsQL encompassed 15 questions relating to the subjects' feelings, social interaction with others, and school. The physical score was derived from answers to 8 questions about the subjects' ease of managing physical activity. Total scores were the sum of all the item scores over the number of items answered on all the scales. Change from baseline values of <0 represents worsening, 0 equals no change, and >0 represents improvement.
Time Frame: Baseline, Month 24
Population: 8 subjects completed the assessment at Month 24.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 8
score on a scale
  Psychosocial Score | 0 [-10 to 28]
  Physical Score | 0 [-19 to 19]
  Total Score | -1.1 [-9 to 25]

7. Secondary Outcome: Change From Baseline to Month 24 in Fabry-Specific Pediatric Health and Pain Questionnaire (FPHPQ) Score for Pain Intensity
Description: The Fabry-specific Pediatric Health and Pain Questionnaire (FPHPQ) included questions about Fabry disease-specific symptoms. The assessment of "How bad is your pain today?" was measured on a 10- point scale from 0 (no pain) to 10 (pain as bad as you can imagine). A decrease from baseline indicates an improvement in the condition.
Time Frame: Baseline, Month 24
Population: 8 subjects completed the FPHPQ pain assessment at Month 24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 8
score on a scale | -1.3 (3.20)

8. Secondary Outcome: Number of Subjects Who Experienced Sudden Onset of Pain As Assessed Using the Fabry-Specific Health and Pain Questionnaire (FPHPQ)
Description: Subjects were asked "In the last 3 months how many times did you experience sudden onset of pain?" and responses were reported in the FPHPQ. Responses were categorized as 0, 1 to 3, 4 to 6, and > 6 occurrences of sudden onset of pain.
Time Frame: Month 24
Population: 8 subjects reported frequency of sudden onset of pain on FPHPQ at Month 24
Measure: Count of Participants; unit: Participants
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 8
Participants
  No occurrences | 3
  1 to 3 occurrences | 4
  4 to 6 occurrences | 0
  >6 occurrences | 1

9. Secondary Outcome: Change From Baseline to Month 24 in Plasma Levels of Lyso-Gb3
Description: Blood samples were collected for measurement of lyso-Gb3 levels in plasma. Plasma levels of lyso-Gb3 were measured using a validated liquid chromatography-mass spectrometry assay.
Time Frame: Baseline, Month 24
Population: 8 subjects had lyso-Gb3 results at Month 24
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 8
ng/mL | 0.05 (1.127)

ADVERSE EVENTS:
Time Frame: Adverse event data collected over duration of the study. Duration of participation varied by patient (range: 181 to 1457 days).
Arm/Group | Migalastat HCl 150 mg
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Migalastat HCl 150 mg (N=16)
Gastroenteritis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Migalastat HCl 150 mg (N=16)
Covid-19 (Infections and infestations) | 3 (6)
Nasopharyngitis (Infections and infestations) | 3 (3)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 1 (1)
Asthenia (General disorders) | 1 (2)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Electrocardiogram T wave biphasic (Investigations) | 1 (1)
Left ventricular mass index (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Paraesthesia (Nervous system disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (2)
Influenza (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (4)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT04049760/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT04049760/SAP_001.pdf